CLINICAL TRIAL: NCT02709265
Title: An Open-Label Phase 1 Study of Aerosolized Amikacin and Fosfomycin Delivered Via the PARI Investigational eFlow Nebulizer System or the PARI LC Sprint Nebulizer in Healthy Volunteers
Brief Title: Open-Label Phase 1 Study of Aerosolized Amikacin and Fosfomycin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardeas Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CAP-01-104
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
MeSH Terms: interventions — Amikacin; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): amikacin/fosfomycin (30/12 mg) delivered via the PARI Investigational eFlow Nebulizer (single dose)
  Interventions: Drug: amikacin/fosfomycin
- Cohort 2 (Experimental): amikacin/fosfomycin (60/24 mg) delivered via the PARI Investigational eFlow Nebulizer (single dose)
  Interventions: Drug: amikacin/fosfomycin
- Cohort 3 (Experimental): amikacin/fosfomycin (90/36 mg) delivered via the PARI Investigational eFlow Nebulizer (single dose)
  Interventions: Drug: amikacin/fosfomycin
- Cohort 4 (Experimental): amikacin/fosfomycin (90/36 mg) delivered via the PARI LC Sprint Nebulizer (single dose)
  Interventions: Drug: amikacin/fosfomycin
- Cohort 5 (Experimental): amikacin/fosfomycin (Dose and Nebulizer to be chosen based on results from Cohorts 1 - 4)
  Interventions: Drug: amikacin/fosfomycin

INTERVENTIONS:
Drug: amikacin/fosfomycin — single aerosolized dose

SUMMARY:
This study will evaluate systemic and urine pharmacokinetics in spontaneously breathing healthy volunteers following a single dose of amikacin/fosfomycin, using the PARI Investigational eFlow Nebulizer System or the PARI LC Sprint Nebulizer. Three doses (30/12 mg, 60/24 mg, 90/36 mg amikacin/fosfomycin) will be evaluated. Following this evaluation, a single dose and nebulizer will be chosen to further evaluate systemic, bronchoalveolar, and urine pharmacokinetics in spontaneously breathing healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1 open-label study of three doses of amikacin/fosfomycin. Approximately 30 healthy volunteers will be dosed in five cohorts of six subjects each. The first (sentinel) subject in each of the first three cohorts will be dosed alone. If no significant safety or tolerability events occur, the remaining five subjects in each of the first three cohorts will be dosed. The first cohort (n=6) will be administered the 30/12 mg dose of amikacin/fosfomycin. The second cohort (n=6) will be administered the 60/24 mg dose of amikacin/fosfomycin. The third cohort (n=6) will be administered the 90/36 mg dose of amikacin/fosfomycin. All doses in cohorts 1, 2, and 3 will be delivered with the PARI Investigational eFlow Nebulizer System. The fourth cohort (n=6) will be administered the 90/36 mg dose of amikacin/fosfomycin using the PARI LC Sprint Nebulizer. The fifth cohort (n=6) will test the lowest dose level at which all subjects achieved > 0.3 µg/mL amikacin peak serum concentration. The nebulizer used to deliver doses in cohort 5 will be determined after amikacin concentrations from cohorts 1 through 4 are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years and ≤ 80 years of age (Cohorts 1, 2, 3, and 4). Males or females aged ≥ 18 years and ≤ 65 years of age (Cohort 5).
* Females of childbearing potential must be using contraception. Acceptable methods of contraception include male or female condom with spermicide gel or foam, hormonal contraceptive combined with a condom, Intrauterine Device (IUD), tubal ligation, diaphragm with spermicide, or total abstinence with a back-up if the subject becomes active.
* Able to communicate with site personnel and to understand and voluntarily sign the Informed Consent Form.

Exclusion Criteria:

* History of previous allergy or sensitivity to amikacin or fosfomycin.
* Use of oral fosfomycin in the 28 days prior to admission to Phase 1 facility.
* History of reactive airways disease (such as asthma or chronic obstructive pulmonary disease [COPD]), cystic fibrosis, or bronchiectasis.
* Human Immunodeficiency Virus (HIV) positive.
* Active Hepatitis B or C.
* Cigarette/e-Cigarette smoking or use of other nicotine or tobacco containing products within seven days prior to study drug administration.
* Positive for drugs of abuse or alcohol use at screening or admission to Phase 1 facility. A Breathalyzer test will be used to screen for the presence of alcohol. A urine standard panel will be used to test for the following substances (with serum testing for confirmation, as needed):

  * Opiates
  * Oxycodone
  * Methadone
  * Cocaine
  * Tetrahydrocannabinol (THC)
  * Benzodiazepines
  * Amphetamines / Methamphetamines
  * Barbiturates
  * Methylenedioxy-methamphetamine (MDMA)
  * Phenylcyclohexyl piperidine (PCP)
  * Tricyclic Antidepressants
* Participation in a clinical study with administration of an investigational drug product within the previous 30 days, or five half-lives of the previously administered investigational product.
* Donation of blood or significant blood loss within the 8 weeks prior to admission to Phase 1 facility.
* Donation of plasma within the week prior to admission to Phase 1 facility.
* Any other condition which in the view of the Investigator is likely to interfere with the study or put the subject at risk.
* Pregnant or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI Investigational eFlow Nebulizer System | 10 minutes to 24 hours post-dose
Peak plasma concentration (Cmax) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI LC Sprint Nebulizer | 10 minutes to 24 hours post-dose

SECONDARY OUTCOMES:
Time to peak plasma concentration (Tmax) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI Investigational eFlow Nebulizer System | 10 minutes to 24 hours post-dose
Time to peak plasma concentration (Tmax) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI LC Sprint Nebulizer | 10 minutes to 24 hours post-dose
Plasma area under the concentration-time curve (AUC) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI Investigational eFlow Nebulizer System | 10 minutes to 24 hours post-dose
Plasma area under the concentration-time curve (AUC) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI LC Sprint Nebulizer | 10 minutes to 24 hours post-dose
Peak bronchoalveolar lavage concentration (Cmax) of amikacin/fosfomycin following delivery of nebulized 30/12 mg, 60/24 mg, or 90/36 mg amikacin/fosfomycin via the PARI Investigational eFlow Nebulizer System or the PARI LC Sprint Nebulizer | 30 minutes post-dose
  The dose and nebulizer used for Cohort 5 will be chosen based on plasma Cmax results from Cohorts 1 - 4.

OTHER OUTCOMES:
Peak urine concentration (Cmax) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI Investigational eFlow Nebulizer System | 0 - 6 hours; 6 - 12 hours; and 12 - 24 hours post-dose
Peak urine concentration (Cmax) of nebulized amikacin/fosfomycin following delivery of 30/12 mg, 60/24 mg, and 90/36 mg amikacin/fosfomycin via the PARI LC Sprint Nebulizer | 0 - 6 hours; 6 - 12 hours; and 12 - 24 hours post-dose
Number of subjects with treatment-related adverse events | 0 - 24 hours post-dose
Change in lung function from pre-dose to post-dose | pre-dose to 15 minutes post-dose
  Spirometry (forced vital capacity, forced expiratory volume in 1 second, and forced expiratory flow in the middle 50% of the exhaled volume) will be measured prior to dosing with study drug and 15 minutes after completing the dose of study drug
Change in vital signs from pre-dose to post-dose | pre-dose to 15 minutes post-dose
  Vital signs (heart rate, respiratory rate, blood pressure, and oximetry) will be measured prior to dosing with study drug and 15 minutes after completing the dose of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No